CLINICAL TRIAL: NCT02740192
Title: Pain Control After Total Knee Arthroplasty: A Prospective, Double-blind Randomized Controlled Trial Examining the Benefit of a Combined Adductor-canal Nerve Block With Periarticular Infiltration Versus Periarticular Injection Alone
Brief Title: Pain Control After Total Knee Arthroplasty: Benefit In Adding Single Shot Adductor Canal Block to Existing Pain Regimen Protocol?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Michael Charters, MD, Staff Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10221
Record Dates: First submitted 2016-03-24; First posted 2016-04-15 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Adductor Canal Block (Experimental): Patients in this group received local infiltration of bupivacaine in the adductor canal after surgery, in addition to the periarticular injection intra-op.
  Interventions: Procedure: Adductor Canal Block; Procedure: Periarticular Injection; Drug: Ropivacaine; Drug: Bupivacaine
- Periarticular Injection (Sham Comparator): Patients in this group received a bandaid at the presumed adductor canal injection site, in addition to the periarticular injection intra-op.
  Interventions: Procedure: Periarticular Injection; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Adductor Canal Block — Post-op adductor canal block using Bupivacaine
  Arms: Adductor Canal Block
Procedure: Periarticular Injection — Intra-op periarticular injection of Ropivacaine
Drug: Ropivacaine — Ropivacaine was used for the periarticular injection
  Other Names: Naropin
Drug: Bupivacaine — Bupivacaine was used for the periarticular injection
  Other Names: Marcaine
  Arms: Adductor Canal Block

SUMMARY:
This is a randomized, double blinded, standard of care controlled clinical trial. All adult patients over eighteen desiring total knee arthroplasty will be eligible. The study compares pain control, opioid consumption, and physical exam findings in patients undergoing total knee arthroplasty between patients receiving adductor canal block and those who receiving periarticular injection alone.

DETAILED DESCRIPTION:
The purpose of this project is to compare the effectiveness of two different but well accepted approaches to nerve blockade in order to improve pain control after total knee arthroplasty. Specifically, this study seeks to identify the if adductor canal blockade provides additional pain relief and decreased morphine consumption when used in addition to a local infiltration of anesthetic (periarticular injection).

Aims:

1. compare pain scores in the post operative period between the two groups.
2. compare morphine equivalent required in the postoperative period
3. compare patient satisfaction with pain control in the post operative period
4. compare physical exam findings such as joint range of motion in the post operative period
5. compare ability to participate with physical therapy in the post operative period

Total knee arthroplasty is associated with intense pain in the post operative period. Pain control is essential in this patient population. Beyond the ethical and humanitarian concerns, pain has been shown in the literature to affect outcomes after total knee replacement. Patients in pain tend to have worse range of motion, decreased participation with physical therapy, increased time to discharge, and downstream medical sequela as well. Pain has been shown to cause or exacerbate delirium in the postoperative period. Patients in pain ambulate less and stay in bed more, therefore increasing the risk of deep vein thrombosis and pulmonary embolism. Patients in pain consume more opioids, which have well known side effects, such as constipation, nausea, vomiting, pruritus, addiction, and altered mental status. Early joint range of motion prevents irreversible joint stiffness and pain, affecting long term outcomes. Pain control in patients undergoing total knee arthroplasty has improved in recent years. The current standard has become a multimodal approach, consisting of preoperative, intraoperative and post operative interventions. The multimodal approach works by preventing or addressing pain at multiple location and targets multiple different pain receptors and pain generators. There has been much attention given to injections and nerve blocks in addition to standard pain medications such as antiinflammatories, acetaminophen, and opioids. There have been many published studies investigating various medication regimens, periarticular injection cocktails, and post operative nerve blocks. These studies have shown that each modality works better than placebo. Several studies have shown that post operative blocks provide additional benefit when used in conjunction with a periarticular injection. These studies were done with femoral nerve catheters and adductor canal catheters that stay in place for several days post operative and require subsequent boluses. No studies in the literature have studied the additional benefit of a single shot adductor canal block. The rationale is that the injection given at the time of surgery should affect the same same local nerves and pain receptors as the adductor canal block, via a different technique. Therefore, the investigators believe the adductor canal block may prove to be of no additional benefit in the investigators patients.

The ultimate goal is identifying the best pain control protocol to decrease pain in the post operative period. Developing this protocol may require the addition or subtraction of various treatment modalities. This study is looking at the adductor canal block, which if found to be unnecessary will prevent patients from receiving unnecessary procedures. If found to be effective at reducing pain, then this study will provide direct evidence for using single shot adductor canal blockade in addition to the periarticular injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 scheduled for primary total knee arthroplasty by four fellowship trained surgeons will be eligible for inclusion.

Exclusion Criteria:

* Patients will be excluded if their medical history presents chronic opioid use (greater than 3 month use),
* pregnancy,
* history of intolerance to medications in the study, and substantial substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Post-operative pain level (Visual Analog Scale) | Through study completion, an average of 3 days
  Patients' pain levels will be recorded every 6 hours using VAS (Visual Analog Scale) by the nursing staff from when the patient arrives on the inpatient floor to when the patient is discharged from the hospital.
Knee flexion and extension Range of Motion (ROM) | Through study completion, an average of 3 days
  Patients' knee ROM will be assessed every morning at 6:30am by the rounding physician on the inpatient floor until the patient is discharged from the hospital.
Distance Walked (meters) | Through study completion, an average of 3 days
  Patients will work with Physical Therapists 2 times day (AM and PM). Distance walked (meters) will be recorded by the Physical Therapist from postoperative day #1 until the patient is discharged from the hospital.
Pain with Ambulation (VAS) | Through study completion, an average of 3 days
  Patients will work with Physical Therapists 2 times day (AM and PM). Pain with ambulation (VAS) will be recorded by the Physical Therapist from postoperative day #1 until the patient is discharged from the hospital.

SECONDARY OUTCOMES:
Pain Medication Intake | Through study completion, an average of 3 days
  Patients' opioid intake (oxycodone, morphine, ms contin, dilaudid, etc) will be calculated and converted to morphine equivalents. The values will be recorded by the rounding physician from when the patient arrives on the inpatient floor to when the patient is discharged from the hospital.
Time to discharge readiness | Through study completion, an average of 3 days
  Time to discharge readiness will be calculated in hours by the rounding physician from when the patient arrives on the inpatient floor to when the patient is discharged from the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States